CLINICAL TRIAL: NCT06495372
Title: Prospective Double-blind Randomized Comparative Study of the Use of Methoxyflurane vs Placebo in the Management of Pain in Oral and Dental Emergencies in Adults: METODO (METhoxyflurane in ODOntology)
Brief Title: Study of the Use of Methoxyflurane vs Placebo in the Management of Pain in Oral and Dental Emergencies in Adults: METODO (METhoxyflurane in ODOntology)
Acronym: METODO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29BRC23.0024 (METODO)
Record Dates: First submitted 2023-12-15; First posted 2024-07-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Dental Pain and Sensation Disorder
MeSH Terms: conditions — Toothache; Sensation Disorders | interventions — Standard of Care; Methoxyflurane; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Experimenta group (standard of care + Methoxyflurane).
- control group (Placebo Comparator)
  Interventions: Drug: control group (standard of care + placebo).

INTERVENTIONS:
Drug: Experimenta group (standard of care + Methoxyflurane). — standard of care + Methoxyflurane
  Arms: Experimental group
Drug: control group (standard of care + placebo). — standard of care + placebo
  Arms: control group

SUMMARY:
With a chronic shortage of dentists in some regions, and an increase in life expectancy and living conditions, the number of patients admitted to oral health emergencies is on the rise. Pain is the main reason for consultation, and is particularly exacerbated in the orofacial sphere. Dental pain has several etiologies: infectious, inflammatory or traumatic accidents.Beyond the ethical aspects of acute pain management, pain relief is a real objective. Despite prioritization systems, patients can wait a long time in an unsettled environment, with tired and sometimes aggressive patients. Numerous recommendations exist to improve analgesia in emergency departments, but there are still difficulties in effectively and rapidly managing acute dental and orofacial pain. To meet this demand and facilitate the treatment process, an alternative solution using methoxyflurane (Penthrox®) could be considered. This product, mainly intended for emergency services, has been approved in Europe since 2016 for the "emergency relief of moderate to severe pain associated with trauma in conscious adult patients". Thus, it would be interesting to assess the value of methoxyflurane (Penthrox®) in the management of pain in oral emergencies as a wait-and-see solution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years)
* Conscious patient consulting an oral emergency department with pain assessed as moderate to severe NRS greater than or equal to 4
* Patient has social security affiliation or who beneficiary of such social security
* Patients who have given informed consent

Exclusion Criteria:

* Patients with a history of allergy to methoxyflurane or any of the components of Penthrox (take into account family history of severe allergic reactions)
* Patients with a history of malignant hyperthermia (known or genetic predisposition)
* Patients with hepatic impairment after use of methoxyflurane or halogenated hydrocarbon anesthesia
* Patients with severe renal Failure
* Patients with altered level of consciousness, whatever the cause: head trauma, drug or alcohol abuse
* Patients with cardiovascular instability or respiratory depression
* Pregnant or breast-feeding patients. Therefore, a urine pregnancy test will be performed for all patients of childbearing age eligible to participate in the study
* Patients under legal protection (guardianship and curatorship) or deprived of liberty
* Patients unable to speak or read French fluently, unable to understand the principle of a numerical scale, anxiety and satisfaction questionnaires, and unable to cooperate with tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by a numerical rating scale at baseline and at T=15min post-treatment | 15 minutes post-treatment
  Pain at baseline and at T=15min post-treatment, measured using a numerical rating scale (NRS) graded from 0 to 10 (0 means no pain, 10 means maximum imaginable pain)

SECONDARY OUTCOMES:
Pain intensity <4/10 (yes/no) at T=15min after treatment | 15 minutes post-treatment
Pain assessed by a numerical rating scale at T=7min (immediate efficacy) | 7 minutes post-treatment
  Pain at T=7 min post-treatment, measured using a numerical rating scale (NRS) graded from 0 to 10 (0 means no pain, 10 means maximum imaginable pain)
Pain assessed by a numerical rating scale at T=40 minutes after treatment and just prior to treatment by the practitioner (persistence of efficacy) | 40 minutes post-treatment
  Pain at T=40 min post-treatment, measured using a numerical rating scale (NRS) graded from 0 to 10 (0 means no pain, 10 means maximum imaginable pain)
Assessment of Anxiety | Just before chairside treatment
  Anxiety, measured at inclusion and just before chairside treatment using a translated and adapted anxiety questionnaire (MDAS: modified dental anxiety scale) Total score is a sum of all five items, range 5 to 25: 5 means not anxious, 25 means extremely anxious
Measuring the amount of local anesthetic used during treatment | 1 day
Post-care satisfaction questionnaire | End of the study (up to 1 day)
  Answers to 4 questions on overall satisfaction of the care, ranging from very dissatisfied to very satisfied
Pain assessed by a numerical rating scale at T=15min according to analgesic associated with methoxyflurane | 15 minutes post-treatment
  Pain at T=15 min post-treatment, measured using a numerical rating scale (NRS) graded from 0 to 10 (0 means no pain, 10 means maximum imaginable pain)
Pain assessed by a numerical rating scale at T=15min according to type of emergency | 15 minutes post-treatment
  Pain at T=15 min post-treatment, measured using a numerical rating scale (NRS) graded from 0 to 10 (0 means no pain, 10 means maximum imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement